CLINICAL TRIAL: NCT00198224
Title: Pilot Study of In Vitro Immunosuppressive Effects of Mycophenolate Mofetil and Valganciclovir in Kidney Transplant Recipients
Brief Title: Immunosuppressive Effects of Mycophenolate Mofetil and Valganciclovir in Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Hoffmann-La Roche (Industry)
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 0212-78; VAL074
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2004-11

CONDITIONS: Renal Failure
Keywords: immunosuppression
MeSH Terms: conditions — Renal Insufficiency | interventions — Phlebotomy

INTERVENTIONS:
Procedure: phlebotomy

SUMMARY:
Valganciclovir (VGCV) has recently been approved by the Food and Drug Administration (FDA) for the treatment and prevention of cytomegalovirus (CMV) retinitis in HIV patients. It is under review for the prevention of CMV disease following organ transplantation. Mycophenolate mofetil (MMF), the morpholinoethyl ester of mycophenolic acid (MPA) is currently the most widespread used immunosuppressant in kidney transplantation. These drugs exerts their effects by blocking the production of DNA primarily in lymphocytes.

Recent studies have suggested that combining both MMF and GCV in vitro may have a beneficial effect on the treatment of CMV infections. However, the effect of these two drugs in combination on the effects of the immune system both in vitro and in vivo have not been studied. Preliminary studies in our lab show that a combination of these two drugs have an additive effect on the level of immunosuppression of both the growth and differentiation of progenitor bone marrow cells as well as lymphocyte proliferation.

This study is designed to test patients degree of immune reactivity both on and off VGCV when used in combination with MMF. Patients will have blood drawn as several time points and an immune assay will be performed to show if VGCV when used in combination with MMF exerts immunosuppressive effects.

DETAILED DESCRIPTION:
Recruitment and screening of subjects will be performed between 4 and 8 weeks after transplantation at which time consent will be obtained. Per clinical standard of care at Indiana University, VGCV is routinely stopped at 12 weeks post transplantation. At week 10 and the day of discontinuation of their prophylaxis the patients will be seen by the study physician. The subjects will also be seen at 2 and 4 weeks after discontinuing VGCV. At each study visit, the subject will have a limited history and physical (H&P) performed, one 3ml light green top (lithium heparin) tube, one 3ml dark green top (sodium heparin) tube, and one 5ml purple top (EDTA) tube will be obtained by phlebotomy during their regularly scheduled blood draw times. This blood will then be used for the Cylex® assay, Flow cytometry and MMF and GCV trough level. The patient's complete blood count and differential as well as drug levels, and medication dosages will be recorded. This information will be used for assure that Cylex® results are not being influenced by changes in immunosuppressive drug levels. The complete blood count and differential will be used to determine absolute neutrophil counts. After the week sixteen visit, the subjects will have completed the protocol. Pregnancy tests will not be performed as patients are not directly receiving any treatment secondary to this study. Flow cytometry will be performed to measure absolute CD4 counts, CD4/CD8 ratios, and look at several activation markers on lymphocytes.

Signed IRB approved informed consent must be obtained from all subjects prior to screening assessments. The following evaluations will be performed prior to initiation of phlebotomy for purposes of this study.

Medical history including age, gender, race, and renal disease, immunosuppressive regimen including dose, level and use of antibody treatment at time of transplant will be noted.

Physical examination including: vital signs, cardiac, and lung evaluation.

Laboratory testing which will be performed as part of standard of care because of the transplant are:

Hematology: complete blood count. Drug level: tacrolimus, cyclosporine and/or sirolimus.

Evaluations during treatment and post treatment

Patients will be followed by surgical co-investigators throughout the entire study.

A limited history and physical examination will be performed as indicated in the schedule of assessments.

Clinical laboratory testing Additional clinical laboratory testing beyond standard of care that will be done for this protocol includes adding a differential to the complete blood count. CBC and drug levels will be noted from already scheduled clinic appointments and post transplant protocols. Research blood levels for GCV and MPA will be run from a 3ml lithium heparin and a 5ml EDTA tube in the research laboratory or at outside laboratory.

Transplant laboratory testing On the testing days an additional 3ml sodium heparin blood tube will be drawn in phlebotomy at the same time the scheduled labs are obtained. Flow cytometric analysis will be performed at times listed above. A 5 tube panel using three color analysis will be performed using approximately 500_L of whole blood from the sodium heparinized tube. The panel will consist of the following staining protocol

Tube 1 - CD 45 FITC / CD 14 PE - Used to locate lymphocyte population as well as determine purity of specimen and monocyte contamination

Tube 2 - _1a FITC/ _1a PE/ _1a PerCP - Isotype control to check for background staining.

Tube 3 - CD 4 FITC/ CD 8 PE / CD 20 PerCP - Used to determine CD4/CD8 ratio as well as determining B cell population counts.

Tube 4 - CD 4 FITC/ CD 25 PE/ HLA - DR PerCP - Check for specific activation markers on CD 4 cells.

Tube 5 - CD 4 FITC/ CD 69 PE/ CD 3 PerCP - Used to get true CD4 counts on T-cells as well as look at another activation marker on CD4 cells.

Cylex immune assay will be run as listed above. This assay requires minimal amount of whole sodium heparinized blood and will be used from same tube as flow analyses. The whole blood is diluted with a saline base diluent. It is then stimulated overnight with phytohemagglutinin. The CD4+ or CD3+ T cells are then isolated using magnetic beads. They are lysed and ATP production is recorded using a luciferase based reaction.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Primary kidney transplant
3. MMF included as part of baseline immunosuppression
4. On valganciclovir for CMV prophylaxis. The dose will vary based on renal function but the standard dose is 900 mg per day
5. No prior episodes of rejection
6. On a stable dose of immunosuppressive medications -

Exclusion Criteria:

1. Previous or multiple transplant patients (e.g. second kidney or simultaneous kidney pancreas patient)
2. Uncontrolled or recurrent infections.
3. Psychiatric disorder -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-01; Study Completion 2005-05

PRIMARY OUTCOMES:
The primary endpoint of this study is the analysis of immune responsiveness in vitro in patients before and after routine cessation of VGCV.

SECONDARY OUTCOMES:
Secondary endpoints of this study are the analysis of absolute neutrophil count before and after routine cessation of VGCV. This will be obtained from the patient's complete blood count and differential.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Pescovitz, MD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University Hospital and Emerson Hall, Indiana University School of Medicine, Indianapolis, Indiana
  - University Hospital, Indianapolis, Indiana